CLINICAL TRIAL: NCT01861678
Title: Randomized Controlled Trial to Evaluate High Tie Versus Low Tie of the Inferior Mesenteric Artery in Rectal Anterior Resection for Rectal Cancer Patients
Brief Title: Randomized Controlled Trial to Evaluate High Tie Versus Low Tie of the Inferior Mesenteric Artery in Anterior Resection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shoichi Fujii, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Shoichi Fujii, MD, PhD, Associate Professor, Yokohama City University Medical Center
Organization: Yokohama City University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YCUMC-D1108013; YokohamaCUMC424 (Other: YokohamaCUMC)
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Rectal Cancer; Colon Rectal Resection
Keywords: Rectal cancer; Anterior resection; High tie of inferior mesenteric artery; Low tie of inferior mesenteric artery; Randomized controlled trial
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High tie of IMA (Active Comparator): In High tie group, IMA was transected at its origin from the abdominal aorta.
  Interventions: Procedure: High tie of IMA
- Low tie of IMA (Experimental): In the low tie of the IMA, IMA was separated after branching to the left colic artery. The lymph node dissection around the IMA at its origin was performed.
  Interventions: Procedure: Low tie of IMA

INTERVENTIONS:
Procedure: High tie of IMA — Conventional technique
  Other Names: High tie
  Arms: High tie of IMA
Procedure: Low tie of IMA — Technique for preserving left colic arterial perfusion
  Other Names: Low tie
  Arms: Low tie of IMA

SUMMARY:
The tying at a radix of the inferior mesenteric artery (IMA) is recognized as radical cure technique in a rectal cancer surgery in Japan. In one side, the preserving the left colic artery (LCA) that is the technique to maintain blood flow of proximal sigmoid colon is performed in practice. However, there is no evidence that shows effectiveness of this technique.

We conducted a randomized trial that compared between high tie and low tie of the IMA in rectal anterior resection to define an appropriate portion of IMA tying.

DETAILED DESCRIPTION:
Patients

* This was a randomized controlled trial conducted at a single institute, which was Yokohama City University Medical Center (Japan).
* 300 patients who underwent anterior resection for rectal cancer were randomly allocated to receive high tie or low tie of the inferior mesenteric artery.

Surgical procedures

* All surgical procedures were performed by one specialized colorectal treatment team. The laparoscopic surgeries were performed by a surgeon who passed the skill accreditation system for laparoscopic gastroenterological surgery was established by the Japanese Society for Endoscopic Surgery (JSES), and all open surgeries were performed under the supervision of these skillful surgeons.
* All operations were performed according to the standard radical cure procedure described in the seventh edition of the Japanese General Rules for Clinical and Pathological Studies on Cancer of the Colon, Rectum and Anus. That is, intestinal excision with lymph node dissection around the IMA at its origin was performed in all surgical procedures. Patients who underwent palliative partial excision were not included.
* In the high tie (HT) of the IMA, IMA was separated at its origin from the abdominal aorta.
* In the low tie (LT) of the IMA, IMA was separated after branching to the left colic artery. The lymph node dissection around the IMA at its origin was performed.

Randomization - To balance the operative backgrounds between HT and LT groups, the patients were stratified by the approach of surgery (open or laparoscopic surgery).

Adjuvant therapy

* When the pathological stage was diagnosed as stage 3 by histological examination of the resected specimen, adjuvant chemotherapy was done with oral fluoropyrimidine anti-cancer drug.
* Neither radiation therapy nor preoperative chemotherapy was given to any patient. Preoperative chemo-radiotherapy even for rectal cancer is not yet standard treatment in Japan.

Assessment parameters

* The preoperative parameters
* Operative assessment parameters
* Postoperative assessment parameters An early postoperative complication was defined as a complication that occurred between the finish of the operation and postoperative day 30. A late postoperative complication was defined as a complication that occurred after postoperative day 30. The terminologies of complications were classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, and grading was done by Classification of Surgical Complication.
* The pathological results were recorded according to the 7th edition of the Japanese General Rules for Clinical and Pathological Studies on Cancer of the Colon, Rectum and Anus and 7th edition of primary tumor, regional nodes, metastasis (TNM) classification. Circumferential margin involvement was defined as exposure of a cancer cell at the vertical dissection surface on histological examination.

Follow-up schedule

- The follow-up schedule was as follows according to stage. Patients with stages 0 and 1 were followed up with outpatient examinations including tumor marker measurements, and chest, abdominal and pelvic computed tomography (CT) once a year for five years. Patients with stage 2 and 3a were examined by CT and tumor marker measurements every six months for the first two years. These examinations were done once a year from the third year to the fifth year. Patients with stage 3b and 3c were examined by CT and tumor marker measurements every four months for the first two years, and every six months from the third year to the fifth year.

Statistical analysis

* The primary endpoint was anastomotic leakage rate.
* The secondary endpoints were operation time, amount of bleeding and 5-year overall survival. To evaluate whether a difference in the operative procedure influences survival including death due to another disease, a comparison of overall survival has meaning. Operation time and amount of bleeding were added to the secondary endpoints because these parameters had a possibility of becoming grounds of selection of the operation method if there were no differences in overall survival.
* A sample size of 284 patients was assured to achieve a power of 70% to detect a difference between the groups using a two-sided Chi-squared test with type I error rate equal to 0.05, when the true complication rates were 4% and 12% for the LT and HT groups, respectively. A sample size of 300 patients was assured to achieve a power of 73% to detect a difference in a same condition. The dropouts were considered and the number of accumulation targets was assumed to be 300 patients to keep a power of more than 70%.
* For continuous variables, data are presented as means ± standard deviation (SD). For categorical variables, data are presented as frequencies and percentages (%). Comparison of the endpoints was based on intention-to-treat principle, that is, the patients who switched to another group during surgery were treated as members of the allocated group. The Chi-squared test was applied to evaluate the significance of differences in proportions, and t-test was used to evaluate the significance of differences in continuous variables. A p-value of less than 0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20 years old or over
* Anterior resection is scheduled for rectal cancer and rectosigmoid cancer preoperatively.
* Histologically proven adenocarcinoma
* Clinical tumor penetrates visceral peritoneum (T4a), no metastasis (M0) or lower T factor
* Elective operation
* Tolerable surgery under general anesthesia
* No history of laparotomy for colorectal resection except appendectomy
* Provided written informed consent

Exclusion Criteria:

* Synchronous or metachronous (within 5 years) malignancy in another organ except carcinoma in situ
* Multiple colorectal cancer that needs reconstruction two or more times
* Acute intestinal obstruction or perforation due to rectal cancer
* Pregnant or lactating women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2006-07; Primary Completion 2012-09 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage rate | 14 days after surgery
  Anastomotic leakage rate is defined as an incontinuity at the anastomosis using circular stapler.

SECONDARY OUTCOMES:
Overall survival | 5 years
  All death is defined as an event of overall survival.
Operation time | 1 day after surgery
Amount of blood loss | 1 day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chikara Kunisaki, Professor, Study Chair — Yokohama City University, Gastroenterological Center
Locations (1):
- Yokohama City University Medical Center, Yokohama, Kanagawa, Japan

REFERENCES:
- [Derived] Fujii S, Ishibe A, Ota M, Watanabe K, Watanabe J, Kunisaki C, Endo I. Randomized clinical trial of high versus low inferior mesenteric artery ligation during anterior resection for rectal cancer. BJS Open. 2018 Jun 8;2(4):195-202. doi: 10.1002/bjs5.71. eCollection 2018 Aug. PMID 30079388